CLINICAL TRIAL: NCT02251951
Title: A Multicenter, Phase II, Single-Arm Clinical Trial of Nab-Paclitaxel as Salvage Treatment for Patients With Locally Advanced or Metastatic Adenocarcinomas of the Stomach and Gastro-esophageal Junction.
Brief Title: Nab-Paclitaxel as Salvage Treatment in Locally Advanced or Metastatic Gastric Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT/12.05
Record Dates: First submitted 2014-07-05; First posted 2014-09-29 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Stomach and Gastro-Esophageal Junction (GEJ) Cancer
Keywords: Cancer; Stomach; Gastro-Esophageal Junction; Salvage treatment; Nab-paclitaxel
MeSH Terms: conditions — Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- nab-Paclitaxel (Experimental): Abraxane
  Interventions: Drug: nab-Paclitaxel

INTERVENTIONS:
Drug: nab-Paclitaxel — Abraxane: 150mg/m2 i.v weekly for 3 consecutive weeks followed by a week of rest (28d)
  Other Names: Abraxane

SUMMARY:
The investigators propose to study the efficacy and safety of nab-Paclitaxel in a Phase II trial of patients with locally advanced or metastatic adenocarcinomas of the stomach and gastro-esophageal junction

DETAILED DESCRIPTION:
Adenocarcinomas of the stomach or gastrointestinal junction refractory/resistant to 1st line chemotherapy are considered as an orphan disease with limited (if any) treatment options. The promising results of Nab-Paclitaxel derived from preclinical studies and from clinical trials conducted in breast cancer patients open the field to develop such therapeutic approaches in other cancers types usually treated with taxanes such as gastric and GEJ adenocarcinomas. We design a phase II study in order to evaluate the effect of nab-Paclitaxel as salvage treatment for patients with advanced cancer of the stomach and GEJ previously treated with the DCF regimen.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old
* Disease progression after treatment with the DCF regimen
* Assessable target lesion(s) as defined by RECIST criteria
* ECOG performance status ≤ 1
* Estimated life expectancy more than 3 months
* Serum bilirubin less than 1.5 times the upper normal limit
* Aspartate Aminotransferase and Alanine Aminotransferase less than 2.5 times the upper normal limit
* Creatinine Clearance ≥50 ml/min
* Neutrophil count more than 1.5x 109 /L
* Platelet count more than 100x 109 /L
* Hemoglobin more than 8g/dL
* Before patient enrollment, written informed consent must be given according to Good Clinical Practice guidelines and national/local regulations.

Exclusion Criteria:

* Gastrointestinal bleeding
* Clinically relevant, symptomatic excessive amounts of ascites resulting in patient's discomfort
* CNS metastases
* Subject pregnant or breast feeding, or planning to become pregnant within 6 months after the end of treatment
* Subject (male or female) is not willing to use highly effective methods of contraception (per institutional standard) during treatment and for 6 months (male or female) after the end of treatment
* Known hypersensitivity reaction to the component of the treatment
* Active infection or malnutrition or bowel obstruction
* Legal incapacity or limited legal capacity
* Definite contraindications for the use of corticosteroids
* History of interstitial lung disease e.g. pneumonitis or pulmonary fibrosis or evidence of interstitial lung disease on baseline chest CT scan
* Chronic inflammation of the bowel
* Clinically significant cardiovascular disease (including myocardial infarction, unstable angina, symptomatic congestive heart failure, serious uncontrolled cardiac arrhythmia) ≤ 1 year before enrollment
* Medical or psychological condition which in the opinion of the investigator would not permit the subject to complete the study or sign meaningful informed consent
* Second primary tumor other than non-melanoma skin cancer or in situ cervical cancer

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-09; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate | Disease evaluation every 8 weeks up to 108 weeks
  Documented response rate will be assessed every two months (8 weeks) until disease progression according to common criteria for tumor response

SECONDARY OUTCOMES:
Disease control rate | Disease evaluation every 8 weeks up to 108 weeks
  Documented disease control rate will be assessed every two months (8 weeks) until disease progression according to common criteria for tumor response
Progression Free Survival | Up to 108 weeks
  From date of randomization until the date of first documented progression or date of death from any cause, whichever come first, assessed up to 108 weeks
Overall Survival | Up to 108 weeks
  From date of randomization until the date of last follow up or death from any cause, assessed up to 108 weeks
Number of Participants with Adverse Events | Every two weeks up to 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: John Souglakos, MD, Principal Investigator — University Hospital of Herklion; Vassilis Georgoulias, MD, Principal Investigator — University Hospital of Heraklion
Locations (6):
- Greece (6):
  - University Hospital of Crete, Dep of Medical Oncology Heraklion, Greece, Heraklion, Crete
  - "Laikon" General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Air Forces Military Hospital of Athens Athens, Greece, Athens
  - SOTIRIA Hospital, Medical Oncology Department, Athens
  - "Ag. Georgios" General Hospital of Chania, Chania
  - "PAPAGEORGIOY" General Hospital of Thessaloniki, Thessaloniki